CLINICAL TRIAL: NCT04986787
Title: Novel, Individualized Brain Stimulation, Network-based Approaches to Improve Cognition in Healthy Seniors and Patients With MCI
Brief Title: Novel, Individualized Brain Stimulation, Network-based Approaches to Improve Cognition
Acronym: NiBS-iCog
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masaryk University (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: GF21-13462L
Record Dates: First submitted 2021-04-19; First posted 2021-08-03 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment; Healthy Aging
Keywords: non-invasive brain stimulation; tACS; TMS; cognition; working memory; MCI; healthy ageing; EEG; neuroimaging (MRI); oscillatory activity
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Entrainment with personalized bi-focal fronto-parietal synchronized tACS in HV - within-frequency (Experimental): double-blind, randomized, sham-controlled, cross-over trials assessing the effects of individualized fronto-parietal tACS on a visual working memory task in aged HV
  Interventions: Device: tACS
- Entrainment with personalized bi-focal fronto-parietal synchronized tACS in HV - cross-frequency (Experimental): double-blind, randomized, sham-controlled, cross-over trials assessing the effects of individualized cross-frequency fronto-parietal tACS stimulation on a visual WM task in aged HV
  Interventions: Device: tACS
- Cerebellar rTMS to modify the effects of cortico-cortical, fronto-parietal tACS in HV (Experimental): double-blind, randomized, sham-controlled, cross-over trial assessing the effects of cerebellar stimulation on individualized fronto-parietal tACS stimulation during a visual WM task in aged HV
  Interventions: Device: tACS; Device: TMS
- Neuromodulation protocol in MCI patients (precise protocol to be chosen on results of previous arms) (Experimental): double-blind, randomized, sham-controlled, cross-over trials assessing the effects of individualized striatal TIS combined with cereberal TMS on a visual working memory task in MCI patients
  Interventions: Device: TMS; Device: TIS

INTERVENTIONS:
Device: tACS — a non-invasive brain stimulation technique that allows interaction with endogenous cortical oscillatory rhythms
  Arms: Cerebellar rTMS to modify the effects of cortico-cortical, fronto-parietal tACS in HV; Entrainment with personalized bi-focal fronto-parietal synchronized tACS in HV - cross-frequency; Entrainment with personalized bi-focal fronto-parietal synchronized tACS in HV - within-frequency
Device: TMS — a noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain, it will be specifically cerebellar stimulation
  Arms: Cerebellar rTMS to modify the effects of cortico-cortical, fronto-parietal tACS in HV; Neuromodulation protocol in MCI patients (precise protocol to be chosen on results of previous arms)
Device: TIS — temporal interference stimulation targeted to striatum, a non-invasive brain stimulation technique that allows interaction with endogenous cortical oscillatory rhythms deep in the brain
  Arms: Neuromodulation protocol in MCI patients (precise protocol to be chosen on results of previous arms)

SUMMARY:
Impaired working memory (WM) plays a crucial role in normal aging, in mild cognitive impairment (MCI) and cognitive decline associated with dementia, such as Alzheimer's disease (AD). The aging-related differences in WM are hypothesized to be based on various neurobiological origins, for example alterations in the dynamic interplay between the large-scale brain networks have proven an important role. Recent studies have shown that non-invasive brain stimulation (NIBS) methods can modulate neuronal activity, plasticity and large-scale brain network interactions. The investigators hypothesize that multifocal NIBS can improve WM. By successive and concurrent stimulation of multiple brain regions of the WM network by transcranial alternating current stimulation (tACS) and/or repetitive transcranial magnetic stimulation (rTMS) the investigators will study dynamic interactions between distinct cortico-cortical and subcortico-cortical brain areas. By leveraging multimodal systems neuroscience information during multifocal stimulation, the investigators expect to acquire better mechanistic understand through which NIBS acts on the brain and improves cognitive functions, such as WM.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) describes an intermediate stage from normal cognitive functioning to dementia, and identifies a spectrum of diseases that includes impairment in both memory and non-memory cognitive domains. A deficient working memory (WM) plays a crucial role in normal aging, MCI, and cognitive decline associated with dementia, such as Alzheimer's disease (AD). WM refers to the on-line temporary storage and manipulation of information to be employed in ongoing processing, and is central to the execution of a variety of daily functions. The loss of WM efficiency related to either aging or neurodegenerative process is hypothesized to have various neurobiological roots, among which altered functioning of the fronto-parietal networks play an important role. The processing, exchange, and storing of information rely on intra- and interregional connectivity that allow neuronal populations to synchronize their firing. Based on this, intra- and cross frequency oscillatory interactions have been demonstrated as core basis for working memory processes, besides other cognitive functions. Any impairment preventing the adaptation and synchronization of the oscillatory activities within this network will inevitably lead to temporary or permanent loss of function.

In this project, based on the mentioned pathophysiological concepts, the investigators will develop and test novel, individualized, multifocal, physiology-inspired non-invasive brain stimulation (NIBS) approaches aimed at enhancing interregional processing in memory-related fronto-parieto-cerebello networks with consecutive behavioral modulation of WM processes impacting on daily life activities in aged healthy volunteers (HV) and MCI patients.

The investigators approach these aims in a step-wise manner: (1) The investigators will explore entrainment of oscillatory activity in the fronto-parietal network with transcranial alternative current stimulation (tACS) at frequencies relevant to memory encoding (theta) to boost WM in healthy seniors. (2) Then, the investigators will explore cross-frequency entrainment of interregional oscillatory interactions in the frontal and parietal target network with bifocal tACS to boost WM in healthy seniors. (3) Based on the current knowledge about the extensive involvement of the cerebellum in cognitive processes by its modulatory effects onto the fronto-parietal networks crucial for cognition, the investigators will leverage our experience in non-invasive modulation of the cerebellar outputs by means of repetitive transcranial magnetic stimulation (rTMS). rTMS over the cerebellum will be applied just before cortical entrainment to further enhance its physiological and behavioral effects. (4) Finally, the investigators will select the most effective approach from the previous work-packages to be applied in MCI patients and quantify the behavioral benefits. Besides the behavioral effects, the investigators will apply multimodal systems neuroscience approaches by means of neuroimaging (structural and functional magnetic resonance imaging; s/fMRI) and electrophysiological (Electroencephalography - EEG, transcranial magnetic stimulation - TMS) methods to determine the underlying network mechanisms and patterns of intrinsic connectivity changes. As there is significant spatial heterogeneity in fronto-parietal peak activity in healthy seniors and patients, stimulation targets will be individually defined based on fMRI. By leveraging the mechanistic aspects derived from individualized multifocal stimulation, the investigators expect to better understand the mechanisms through which NIBS techniques act on the brain and improve cognitive functions. The investigators will also test and quantify within a virtual reality (VR) task how well the intervention-driven cognitive improvement translates into daily life.

ELIGIBILITY:
Inclusion Criteria:

* normal cognitive performance as assessed by a cognitive screening for healthy subjects
* mild cognitive impairment as assessed by detailed cognitive testing ± positive AD diagnostic biomarkers for MCI subjects

Exclusion Criteria:

* Psychiatric disorders including major depression, major vascular lesions, or other brain pathologies that might present with cognitive decline.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Working memory performance | through study completion, an average of 1 year
  We will compare the baseline-normalized reaction time and error rate of a N-back task between the real and sham stimulation condition in a cross-over design.

SECONDARY OUTCOMES:
The reproducibility of the outcomes of this proof-of-concept brain stimulation in MCI between centers | through study completion, an average of 1 year
  Twenty MCI patients will be recruited in each participating center. The reproducibility of the effects induced by the intervention will be assessed by comparing the baseline-normalized error rate of a N-back task between the two centers.
The neural underpinning of NIBS-induced changes quantified by s/fMRI and network-based analytical approaches. | The changes will be computed from the difference between connectivity at baseline and 1 hour post-stimulation.
  The changes in intra- and inter-regional fMRI connectivity within and between cognitive brain networks will be compared between the real and sham stimulations.
The neural underpinning of NIBS-induced changes quantified by EEG. | Baseline and 1 hour after the delivery of real or sham intervention - cross-over design.
  We will measure cortical excitability by TMS-EEG pairing via TMS-evoked potentials.
Transfer of the acquired WM abilities during the intervention into a daily-life relevant scenario as assessed by The Virtual Supermarket Shopping Task. | through study completion, an average of 1 year
  The accuracy of the post-stimulation WM task in a VR-based daily life scenario as assessed by The Virtual Supermarket Shopping Task will be compared between the real or sham intervention (cross-over design).

CONTACTS AND LOCATIONS:
Overall Officials: Friedhelm C. Hummel, Principal Investigator — Ecole Polytechnique Fédérale de Lausanne; Irena Rektorova, Principal Investigator — CEITEC Masaryk University
Locations (1):
- Ceitec Masaryk University, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No
Data will be shared only within both centres

REFERENCES:
- [Background] Saunders NL, Summers MJ. Attention and working memory deficits in mild cognitive impairment. J Clin Exp Neuropsychol. 2010 Apr;32(4):350-7. doi: 10.1080/13803390903042379. Epub 2009 Sep 25. PMID 19787522
- [Background] Johnson EL, Dewar CD, Solbakk AK, Endestad T, Meling TR, Knight RT. Bidirectional Frontoparietal Oscillatory Systems Support Working Memory. Curr Biol. 2017 Jun 19;27(12):1829-1835.e4. doi: 10.1016/j.cub.2017.05.046. Epub 2017 Jun 9. PMID 28602658
- [Background] Roux F, Uhlhaas PJ. Working memory and neural oscillations: alpha-gamma versus theta-gamma codes for distinct WM information? Trends Cogn Sci. 2014 Jan;18(1):16-25. doi: 10.1016/j.tics.2013.10.010. Epub 2013 Nov 19. PMID 24268290
- [Background] Kornblith S, Buschman TJ, Miller EK. Stimulus Load and Oscillatory Activity in Higher Cortex. Cereb Cortex. 2016 Sep;26(9):3772-84. doi: 10.1093/cercor/bhv182. Epub 2015 Aug 18. PMID 26286916
- [Background] Eldaief MC, Halko MA, Buckner RL, Pascual-Leone A. Transcranial magnetic stimulation modulates the brain's intrinsic activity in a frequency-dependent manner. Proc Natl Acad Sci U S A. 2011 Dec 27;108(52):21229-34. doi: 10.1073/pnas.1113103109. Epub 2011 Dec 12. PMID 22160708
- [Background] Anderkova L, Pizem D, Klobusiakova P, Gajdos M, Koritakova E, Rektorova I. Theta Burst Stimulation Enhances Connectivity of the Dorsal Attention Network in Young Healthy Subjects: An Exploratory Study. Neural Plast. 2018 Mar 13;2018:3106918. doi: 10.1155/2018/3106918. eCollection 2018. PMID 29725346
- [Background] Novakova L, Gajdos M, Rektorova I. Theta-burst transcranial magnetic stimulation induced cognitive task-related decrease in activity of default mode network: An exploratory study. Brain Stimul. 2020 May-Jun;13(3):597-599. doi: 10.1016/j.brs.2020.01.015. Epub 2020 Jan 31. No abstract available. PMID 32289683
- [Background] Plechata A, Sahula V, Fayette D, Fajnerova I. Age-Related Differences With Immersive and Non-immersive Virtual Reality in Memory Assessment. Front Psychol. 2019 Jun 11;10:1330. doi: 10.3389/fpsyg.2019.01330. eCollection 2019. PMID 31244729